CLINICAL TRIAL: NCT00470561
Title: The Effect of Aspirin on Mammogram Density (TEAM)
Brief Title: Effect of Aspirin on Mammogram Density in Healthy Postmenopausal Women With a Moderate or High Level of Breast Density
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Anne McTiernan, MD PhD, FHCRC
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: PHS 1908.00; FHCRC-PHS-1908.00; FHCRC-1908; CDR0000544639 (Registry Identifier: PDQ); NCT00464906 (obsolete NCT alias)
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-11

CONDITIONS: Mammographic Breast Density
Keywords: mammographic breast density aspirin
MeSH Terms: interventions — Aspirin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin (Active Comparator)
  Interventions: Drug: Aspirin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — Two 325 mg doses of aspirin per day for 6 months
  Other Names: Acetylsalicylic acid
  Arms: Aspirin
Drug: Placebo — Two placebo pills per day for 6 months
  Other Names: Placebo, sugar pill
  Arms: Placebo

SUMMARY:
RATIONALE: Aspirin may be effective in reducing breast density in healthy postmenopausal women with a moderate or high level of breast density.

PURPOSE: This randomized clinical trial is studying the effect of aspirin on mammogram density compared with a placebo in healthy postmenopausal women with a moderate or high level of breast density.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the effect of acetylsalicylic acid (aspirin) vs placebo on mammographic density in healthy postmenopausal women with a moderate or high level of breast density.

Secondary

* Determine whether there is a differential response in mammogram density to aspirin treatments in individual homozygous wild-type, heterozygous, and homozygous variant for several UGT gene polymorphisms.
* Determine the effect of aspirin therapy on potential adverse events, including gastrointestinal symptoms and signs, bleeding events, blood pressure, and other major comorbidities and hospitalizations, as well as generalized symptoms, in these participants.
* Determine the effects of aspirin therapy on putative biomarkers of breast and ovarian cancer that are currently being validated as part of ongoing Fred Hutchinson Cancer Research Center Ovarian SPORE activities.
* Determine the effects of aspirin therapy on levels of serum estradiol, estrone and sex hormone binding globulin (SHBG) as measured by radioimmunoassay at baseline and 6 month timepoints

OUTLINE: This is a randomized, placebo-controlled, double-blind study. Participants are randomized to 1 of 2 treatment arms.

* Arm I: Participants receive oral acetylsalicylic acid (aspirin) daily for 6 months.
* Arm II: Participants receive oral placebo daily for 6 months. In both arms, participants undergo a repeat mammogram at 6 months.

Blood and urine samples are collected at baseline and at 6 months. Single-nucleotide polymorphisms in the UGT genes and variable number of tandem repeat-type polymorphisms are genotyped.

PROJECTED ACCRUAL: A total of 144 participants will be accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA:

* Moderate or high density breast tissue on mammogram within the past 4 months

  * Breast Imaging-Reporting and Data System (BIRAD) class 2-4 or digitized mammogram with ≥ 25% density
* Healthy without serious comorbidities
* Female
* Postmenopausal
* More than 3 weeks since prior and no other concurrent use (2 or more times per week) of acetylsalicylic acid (aspirin), ibuprofen, or other NSAIDs

EXCLUSION CRITERIA:

* history of breast cancer, including ductal carcinoma in situ or lobular carcinoma in situ
* history of illness for which NSAIDs are typically primary therapy (e.g., rheumatoid arthritis)
* Allergy to NSAIDs
* Anemia (hematocrit < 35%), abnormal bleeding tests, or bleeding disorders
* Gastrointestinal (GI) ulcer or history of GI bleeding
* Adverse reactions to aspirin acid or other NSAIDs
* Renal disease
* Asthma
* Current or chronic liver disease
* History of hemorrhagic stroke or transient ischemic attack
* History of coronary artery disease, including any of the following:

  * Myocardial infarction (MI)
  * Angina
  * Coronary artery disease documented on cardiac catheterization, exercise thallium, or exercise echocardiogram
* Strong family history of coronary artery disease (i.e., mother with MI before 55 years of age, father with MI before 45 years of age)
* Documented carotid artery disease
* Diabetes
* Uncontrolled hypertension
* No planned extensive weight loss in the next 6 months (≥ 10 pounds)
* More than 2 alcoholic drinks daily
* Mental illness or alcohol or drug abuse
* Prior angioplasty or coronary artery bypass grafting
* Prior breast implantation or reduction surgery
* Less than 6 months since prior hormones for menopause (including pills, patches, vaginal route), tamoxifen citrate, raloxifene, other hormonal therapy, or herbal or soy preparations
* Concurrent anticoagulation medication

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2005-11; Primary Completion 2007-06 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Comparison of the effect of acetylsalicylic acid (aspirin) vs placebo on mammographic density | Baseline and end-of-study (6 month timepoint)

SECONDARY OUTCOMES:
Differential response in mammogram density to aspirin treatments in individual homozygous wild-type, heterozygous, and homozygous variant for several UGT gene polymorphisms | Baseline and end-of-study (6 month timepoint)
  Changes at baseline and 6 month timepoint in mammographic density; measurements of single numcleotide polymorphisms in specific genes from a single DNA samples
Adverse events | Collected over the course of tehestudy
Putative biomarkers of breast and ovarian cancer | Baseline and end-of-study (6 month timepoint)
Comparison of the effect of aspiring vs placebo on serum levels of estradiol, estrone and sex hormone binding globulin | Baseline and 6 month timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Urban, ScD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States